CLINICAL TRIAL: NCT00519675
Title: Open Label Treatment of Patients With Chronic Hand Dermatitis Who Have Participated in a Previous Clinical Trial Involving Oral Alitretinoin
Brief Title: Alitretinoin in the Treatment of Chronic Hand Eczema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAP00731
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Eczema
Keywords: Chronic hand eczema; Chronic hand dermatitis; Patients with chronic hand eczema, who are refractory to topical corticosteroids
MeSH Terms: conditions — Eczema | interventions — Alitretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: alitretinoin

SUMMARY:
The purpose of the study is to investigate the safety and efficacy of alitretinoin in chronic hand eczema that is refractory to topical corticosteroids.

DETAILED DESCRIPTION:
Chronic hand eczema is a frequent and distressing disease. The course of the disease is of chronic-relapsing nature. In a phase III study alitretinoin was clinically effective for patients with severe chronic hand eczema refractory to topical treatment. This study investigates the safety and efficacy of alitretinoin who previously have participated in a clinical trial involving alitretinoin.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in therapeutic trials involving chronic hand eczema
* Relapse of chronic hand eczema, defined as 75% of the baseline initial total lesion symptom score

Exclusion Criteria:

* Patients whose disease is adequately controlled by standard non-medicated skin care and topical corticosteroid therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
Safety assessments

SECONDARY OUTCOMES:
Efficacy (Physicians Global Assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Maares, MD, Study Director — Basilea Pharmaceutica
Locations (4):
- France (2):
  - Paris
  - Saint-Etienne
- Germany (2):
  - Berlin
  - Dresden